CLINICAL TRIAL: NCT00751660
Title: Early Detection of Lung Cancer - A Pan Canadian Study
Brief Title: Screening Methods in Finding Lung Cancer Early in Current or Former Smokers
Acronym: Pan Can
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000598586; BCCA-H08-01132
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Tobacco Use Disorder
Keywords: small cell lung cancer; non-small cell lung cancer; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: screening questionnaire administration
Procedure: bronchoscopic and lung imaging studies
Procedure: computed tomography
Procedure: endoscopic biopsy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Screening may help doctors find lung cancer sooner, when it may be easier to treat.

PURPOSE: This clinical trial is studying screening methods to see how well they find lung cancer early in current or former smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a new multi-modal screening strategy and integrated methods to detect lung cancer early in current and former smokers.
* To evaluate the impact of the screening modalities on the quality of life of these participants.
* To develop a decision analytic framework for determining the cost and effectiveness of a novel lung cancer screening strategy in Canada.

OUTLINE: This is a multicenter study.

Participants undergo spirometry at baseline. Participants also undergo spiral CT scan at baseline and then at 1 and 2 years. Participants with semi-solid or solid nodules of 5-10 mm or ground glass opacity (GGO) 8-10 mm or those with growth of an existing nodule, development of a solid component in GGO, or a new nodule undergo an additional CT scan at 3 months. Some participants also undergo autofluorescence and white light bronchoscopy and bronchial biopsies.

Blood samples are collected at baseline and then annually for 2 years for biomarker studies. Participants diagnosed with lung cancer undergo additional blood sample collection for biomarker studies.

Participants complete questionnaires on sociodemographic factors, smoking, occupational exposure, family history, medical data, quality of life, and anxiety at baseline and then every 6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current or former smoker

  * A former smoker is defined as one who has stopped smoking ≥ 1 year but < 15 years ago
* Estimated 1-year lung cancer risk ≥ 1%

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Not pregnant
* Willing to undergo a spiral chest CT scan
* No severe heart disease (e.g., unstable angina or chronic congestive heart failure)
* No acute or chronic respiratory failure
* No bleeding disorder
* No other medical condition that, in the opinion of the investigator, would preclude the participant's safety during study participation or that would unlikely benefit the participant from screening due to shortened life expectancy from the co-morbidity
* No diagnosis of cancer, except for any of the following that were previously treated ≥ 5 years ago:

  * Non-melanomatous skin cancer
  * Localized prostate cancer
  * Carcinoma in situ of the cervix
  * Superficial bladder cancer
* No known reaction to xylocaine, salbutamol, midazolam, or alfentanil

PRIOR CONCURRENT THERAPY:

* More than 2 years since prior chest CT scan
* No concurrent anti-coagulant treatment (e.g., warfarin or heparin)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2504 (Actual)
Dates: Start 2008-09; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Number of lung cancer cases detected early by spiral CT scan and autofluorescence bronchoscopy | 24 months
Number of interval lung cancer cases | 60 months

SECONDARY OUTCOMES:
Stage distribution of lung cancer cases | 60 months
Prevalence of lung nodules and differences in geographic distribution across Canada | 60 months
Rate of detection of other incidental significant treatable diseases | 60 months
Type and costs of downstream investigation and treatment related to abnormalities found by the screening procedures, whether the final diagnosis is lung cancer or not | 60 months
Potential physical and psychosocial impact on participants | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Principal Investigator — British Columbia Cancer Agency
Locations (6):
- Canada (6):
  - University of Calgary Health Sciences Centre, Calgary, Alberta
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - L'Hopital Laval, Québec, Quebec

REFERENCES:
- [Derived] Goffin JR, Pond GR, Puksa S, Tremblay A, Johnston M, Goss G, Nicholas G, Martel S, Bhatia R, Liu G, Schmidt H, Atkar-Khattra S, McWilliams A, Tsao MS, Tammemagi MC, Lam S. Chronic obstructive pulmonary disease prevalence and prediction in a high-risk lung cancer screening population. BMC Pulm Med. 2020 Nov 16;20(1):300. doi: 10.1186/s12890-020-01344-y. PMID 33198781
- [Derived] Rudkowski JL, Pond GR, Tremblay A, Johnston M, Goss G, Nicholas G, Martel S, Bhatia R, Liu G, Schmidt H, Tammemagi MC, Atkar-Khattra S, Tsao MS, Lam S, Goffin JR. Trial marketing in the Pan-Canadian Early Detection of Lung Cancer Study. Clin Trials. 2020 Apr;17(2):202-211. doi: 10.1177/1740774519895966. Epub 2020 Jan 2. PMID 31894702
- [Derived] Taghizadeh N, Tremblay A, Cressman S, Peacock S, McWilliams AM, MacEachern P, Johnston MR, Goffin J, Goss G, Nicholas G, Martel S, Laberge F, Bhatia R, Liu G, Schmidt H, Atkar-Khattra S, Tsao MS, Tammemagi MC, Lam SC; Pan-Canadian Early Lung Cancer Study Group. Health-related quality of life and anxiety in the PAN-CAN lung cancer screening cohort. BMJ Open. 2019 Jan 17;9(1):e024719. doi: 10.1136/bmjopen-2018-024719. PMID 30659040
- [Derived] Tammemagi MC, Schmidt H, Martel S, McWilliams A, Goffin JR, Johnston MR, Nicholas G, Tremblay A, Bhatia R, Liu G, Soghrati K, Yasufuku K, Hwang DM, Laberge F, Gingras M, Pasian S, Couture C, Mayo JR, Nasute Fauerbach PV, Atkar-Khattra S, Peacock SJ, Cressman S, Ionescu D, English JC, Finley RJ, Yee J, Puksa S, Stewart L, Tsai S, Haider E, Boylan C, Cutz JC, Manos D, Xu Z, Goss GD, Seely JM, Amjadi K, Sekhon HS, Burrowes P, MacEachern P, Urbanski S, Sin DD, Tan WC, Leighl NB, Shepherd FA, Evans WK, Tsao MS, Lam S; PanCan Study Team. Participant selection for lung cancer screening by risk modelling (the Pan-Canadian Early Detection of Lung Cancer [PanCan] study): a single-arm, prospective study. Lancet Oncol. 2017 Nov;18(11):1523-1531. doi: 10.1016/S1470-2045(17)30597-1. Epub 2017 Oct 18. PMID 29055736
- [Derived] Zafari Z, Sin DD, Postma DS, Lofdahl CG, Vonk J, Bryan S, Lam S, Tammemagi CM, Khakban R, Man SFP, Tashkin D, Wise RA, Connett JE, McManus B, Ng R, Hollander Z, Sadatsafavi M. Individualized prediction of lung-function decline in chronic obstructive pulmonary disease. CMAJ. 2016 Oct 4;188(14):1004-1011. doi: 10.1503/cmaj.151483. Epub 2016 Aug 2. PMID 27486205
- [Derived] Tremblay A, Taghizadeh N, McWilliams AM, MacEachern P, Stather DR, Soghrati K, Puksa S, Goffin JR, Yasufuku K, Amjadi K, Nicholas G, Martel S, Laberge F, Johnston M, Shepherd FA, Ionescu DN, Urbanski S, Hwang D, Cutz JC, Sekhon HS, Couture C, Xu Z, Sutedja TG, Atkar-Khattra S, Tammemagi MC, Tsao MS, Lam SC; Pan-Canadian Early Lung Cancer Study Group. Low Prevalence of High-Grade Lesions Detected With Autofluorescence Bronchoscopy in the Setting of Lung Cancer Screening in the Pan-Canadian Lung Cancer Screening Study. Chest. 2016 Nov;150(5):1015-1022. doi: 10.1016/j.chest.2016.04.019. Epub 2016 Apr 30. PMID 27142184
- [Derived] McWilliams A, Tammemagi MC, Mayo JR, Roberts H, Liu G, Soghrati K, Yasufuku K, Martel S, Laberge F, Gingras M, Atkar-Khattra S, Berg CD, Evans K, Finley R, Yee J, English J, Nasute P, Goffin J, Puksa S, Stewart L, Tsai S, Johnston MR, Manos D, Nicholas G, Goss GD, Seely JM, Amjadi K, Tremblay A, Burrowes P, MacEachern P, Bhatia R, Tsao MS, Lam S. Probability of cancer in pulmonary nodules detected on first screening CT. N Engl J Med. 2013 Sep 5;369(10):910-9. doi: 10.1056/NEJMoa1214726. PMID 24004118